CLINICAL TRIAL: NCT00400491
Title: Vitamin D Supplementation to Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Tromso (Other)
Responsible Party: Professor Roy Bremnes, University of Tromso
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EUDRACT-2006-000177-30
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2008-05

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; insulin; glycated hemoglobin; cholecalciferol; vitamin D
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Cholecalciferol (vitamin D)
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cholecalciferol (vitamin D) — Cholecalciferol capsule 20.000 IU twice per week for 6 months
  Other Names: vitamin D
  Arms: 1
Drug: Placebo — Placebo capsule twice a week, identical to the cholecalciferol capsules
  Arms: 2

SUMMARY:
The purpose of the study is to evaluate if supplementation with vitamin D in a dose of 40.000 IU per week will result in improved metabolic control in patients with type 2 diabetes.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate if supplementation with vitamin D in a dose of 40.000 IU per week will result in improved metabolic control in patients with type 2 diabetes.

We will include 70 patients with type 2 diabetes. They will be treated with 40.000 IU cholecalciferol per week (or placebo) for 6 months. Metabolic control will be evaluated with measurements of glycated hemoglobin, home glucose measurements, and fasting blod glucose and serum insulin. Only subjects using insulin at bedtime combined with metformin during the day will be included.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 1 year
* age 21-75 years
* long-acting insulin at bedtime
* metformin during the day
* for women of child bearing age use of reliable method of birth control

Exclusion Criteria:

* serum creatinine above 130 umol/l for men and above 110 for women
* systolic blood pressure > 175 or diastolic > 104 mmHg
* heart disease
* serum calcium > 2.54 mmol/l
* history of renal stones

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-06; Primary Completion 2007-08 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
glycated hemoglobin | 6 months

SECONDARY OUTCOMES:
blood pressure | 6 months
body weight | 6 months
Hip/waist ratio | 6 months
lipids | 6 months
Hs-CRP | 6 months
insulin sensitivity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Jorde, Professor, Principal Investigator — University of Tromsø, Tromsø
Locations (1):
- Clinical Research Unit, University Hospital of North Norway, Tromsø, Tromsø, Norway